CLINICAL TRIAL: NCT03415542
Title: When Outcomes Matter: A Temporal Analysis of Instrumental and Affective Outcomes of Exercise Behavior Using Ecological Momentary Assessment
Brief Title: A Comparison of Exercise Beliefs to Same-day Exercise Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1604001464
Record Dates: First submitted 2017-12-06; First posted 2018-01-30 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Exercise
Keywords: Attitudes; Ecological momentary assessment
MeSH Terms: conditions — Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Other): Participants receive a print-based exercise promotion program across 12 weeks and are asked to monitor their exercise behavior using an app on their cell phone.
  Interventions: Behavioral: Exercise Promotion

INTERVENTIONS:
Behavioral: Exercise Promotion — Evidence-based techniques (goal-setting, reduced barriers) for increasing exercise behavior

SUMMARY:
Regular aerobic exercise is associated with reduced risk of multiple cancers, yet the majority of adults are inactive. Across health behavior theories, the expectations people have about the outcomes of exercise influence their decision to exercise. Extending prior work, a fine-grained analysis of the relationship between perceived outcomes and daily exercise behavior will be achieved using ecological momentary assessment methods to measure perceived outcomes, and accelerometry to measure exercise objectively. The results of this research will inform exercise promotion efforts by determining how perceptions and temporal factors interact to predict exercise behavior.

DETAILED DESCRIPTION:
There is strong evidence for an association between regular physical activity and reduced risk for cancers of the breast and colon. The majority of adults do not engage in enough physical activity. Motivating adults to exercise is critical to cancer prevention efforts. However, additional work is needed to improve the theoretical frameworks applied to exercise promotion. The most often cited theories of health promotion include the outcomes of a target behavior as important determinants. The perceptions people have about the outcomes of exercise, and more generally attitudes about exercise, are associated with exercise participation. Conceptualizations of perceived outcomes are categorized by whether they are instrumental (i.e. utility-based) or affective (i.e. feeling-based) in nature. Recent efforts to compare the relative predictive power of instrumental and affective attitudes suggest that affective attitudes may better predict exercise behavior. Aim 1 of this proposal seeks to compare the relative influence of instrumental versus affective attitudes on exercise behavior. Another distinction can be made between perceptions that are held temporally proximal versus distal to exercise behavior. In the vast majority of relevant research in the exercise field, perceptions are assessed and then future exercise behavior is assessed months later via self-report. However, day to day perceptions and exercise behavior is largely unknown. The temporal distance of perceptions from the decision to exercise can be significantly shortened using ecological momentary assessments. Aim 2 of this proposal seeks to compare the relative predictive power of temporally distal versus proximal perceptions on exercise behavior. Finally, aim 3 will examine the interaction between instrumental/affective and temporally proximal/distal attitudes for predicting exercise behavior. The proposed research seeks to contribute to cancer prevention efforts by examining underlying perceptions that motivate the day to day decision to exercise. In particular, technological advances in mobile platforms to deliver interventions to people wherever they are requires better support for how to apply these methods. Using theory-based, empirically supported concepts, this longitudinal study will follow previously inactive adults over 12 weeks using electronic diaries to measure their perceptions and exercise behavior change while they receive an exercise intervention. This study will provide a fine-grained examination of the determinants of exercise targeted in exercise promotion interventions. The results will inform future efforts to promote exercise using mobile technologies by determining what types of beliefs (instrumental/affective) and what times (temporal proximity to behavior) are most critical times to intervene.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, inactive adults 18-65

Exclusion Criteria:

* Chronic diseases, recent hospitalization for mental health problems, binge drinking, physical limitations that would make exercise unsafe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Exercise behavior | 1 day
  Examine the association between attitudes and exercise behavior defined by the time of the start and end of each exercise session

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Emerson, MS, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Upon request, data may be shared with other researchers